CLINICAL TRIAL: NCT04074278
Title: Novel Equations for Estimating Lean Body Mass in Patients With Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong Jie, Clinical Professor of Institute of Nephrology, Division of Renal, Peking University First Hospital
Other Study IDs: LBM eqations
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Lean Body Mass; Chronic Kidney Diseases
Keywords: mid-arm muscle circumference; handgrip strength; dual-energy x-ray absorptiometry
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- development groups: The development groups included 150 patients derived from outpatients in Peking University First Hospital, between March 1st, 2014 and November 26th 2014.
- validation groups: The validation groups included 150 patients derived from outpatients in Peking University First Hospital, between November 27th 2014 and December 1st, 2015.

SUMMARY:
Simplified methods to estimate lean body mass (LBM), an important nutritional measure representing muscle mass and somatic protein, are lacking in non-dialyzed patients with chronic kidney disease (CKD).

Objective: We developed and tested a reliable equations for estimation of LBM in daily clinical practice.

DETAILED DESCRIPTION:
Two cross-sectional data sets were derived from outpatients with CKD stage 3-5 in Peking University First Hospital.Two equations for estimating LBM based on midarm muscle circumference (MAMC) or hand grip strength (HGS)were developed and validated in CKD patients with dual-energy x-ray absorptiometry (DEXA) as referenced gold method. Demographic data, comorbidity, and other clinical variables were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* non-dialyzed patients with CKD stage 3-5
* clinical stable
* a willingness to be examined with all measurements being taken simultaneously.

Exclusion Criteria:

* systemic infections, acute cardiovascular events, operations, trauma, active hepatitis or tumor
* severe edema within one month prior to the study
* chronic infections, connective tissue disease, hyper- or hypothyroidism, amputations or pregnancy,
* taking immunosuppressive agents and anti-inflammatory medication chronically

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The development and validation groups both included 150 non-dialyzed patients with CKD stage 3-5.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
LBM_DEXA | between March 1st, 2014 and December 1st, 2015
  lean body mass measured by dual-energy x-ray absorptiometry (DEXA)

CONTACTS AND LOCATIONS:
Locations (1):
- Renal Division and Institute of Nephrology, Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No